CLINICAL TRIAL: NCT07360002
Title: The Randomized Controlled Study of Shenqi Yishen Granules in the Treatment of IgA Nephropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keda Lu (Other)
Collaborators: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); The Second Affiliated Hospital of Zhejiang Chinese Medical University (Other); Red Cross Hospital, Hangzhou, China (Other); Hangzhou Traditional Chinese Medicine Hospital (Unknown); Zhenhai District Traditional Chinese Medicine Hospital (Unknown); Jiangsu Provincial Hospital of Traditional Chinese Medicine (Unknown); Shao Yifu Hospital of Zhejiang Medical University (Unknown); Hangzhou First People's Hospital, School of Medicine, Zhejiang Universiry (Unknown); Yuyao City Traditional Chinese Medicine Hospital (Unknown); First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine (Unknown); Affiliated Hospital of Jiaxing University (Other); Hangzhou Xiaoshan First People's Hospital (Unknown); Shanghai 6th People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Keda Lu, Professor, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZSLL-KY-2025-129-01
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: IgA Nephropathy (IgAN)
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Shenqi Yishen Granules + Irbesartan
  Interventions: Drug: Shenqi Yishen Granules
- Control Group (Placebo Comparator): Chinese herbal placebo + Irbesartan
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Shenqi Yishen Granules — A traditional Chinese medicine compound for the treatment of IgA nephropathy
  Other Names: Irbesartan
  Arms: Treatment group
Drug: Placebo — a look-alike substance that contains no drug
  Other Names: Irbesartan
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to learn if Shenqi Yishen Granules works to treat IgA Nephropathy in adults. It will also learn about the safety of Shenqi Yishen Granules. The main questions it aims to answer are:

Does Shenqi Yishen Granules lower 24-hour urinary protein quantification of participants? What medical problems do participants have when taking Shenqi Yishen Granules? Researchers will compare Shenqi Yishen Granules to a placebo (a look-alike substance that contains no drug) to see if Shenqi Yishen Granules works to treat IgA Nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for IgA nephropathy and CKD stages 1-2, 24h-HPro > 0.3g;
2. Meets the diagnostic criteria for "qi and yin deficiency syndrome" according to Traditional Chinese Medicine;
3. Age between 18 and 75 years, gender;
4. Infection, acidosis, electrolyte imbalance, hypertension, etc., are well controlled;
5. No failure of other organ functions;
6. Have good compliance, have not participated in other clinical trials in the past six months; are informed and voluntarily willing to participate in the clinical study.

Exclusion Criteria:

* (1) Immediate dialysis treatment is required; currently undergoing treatment with hormones, non-steroidal anti-inflammatory drugs, or immunosuppressive agents; (2) Patients with acute infectious diseases or those under surgical or traumatic stress; (3) Patients with chronic infectious diseases such as active chronic hepatitis B,, decompensated cirrhosis, or active tuberculosis; (4) Patients with severe organ dysfunction affecting survival, such as malignant tumors or HIV infection; (5) Patients with severe primary diseases of the cardiovascular, hematological, neurological, digestive, or respiratory systems, or those with a significant tendency to bleed; (6) Patients with life-threatening conditions such as hyperkalemia or heart failure; (7) Patients with a GFR fluctuation of ≥30% within the past 3 months; (8) Patients with severe allergies to certain known drugs in this study or unable to tolerate them; (9) Patients who are pregnant or breastfeeding; (10) Patients with a history of drug abuse or who have used immunosuppressive agents or glucocorticoids in the past 3 months; (11) Patients with major bleeding or blood transfusion history in the past 3 months, or those with severe clinical infections or signs of acidosis; (12) Patients currently participating in other clinical trials or undergoing other Chinese herbal treatments that may affect efficacy assessment; (13) Patients planning or having undergone kidney transplantation, or those with acute or chronic kidney failure requiring immediate replacement therapy; (14) Patients with post-renal factors, such as obstruction (including stones, uric acid crystals, or tumors) causing acute kidney injury; (15) Patients with a history of mental illness or communication/cognitive impairments leading to poor compliance and inability to cooperate; (16) Non-Asian individuals.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
24-hour urinary protein quantification | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  24-hour urinary protein quantification
Protein-to-creatinine rati | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  Concentration of Protein-to-creatinine rati

SECONDARY OUTCOMES:
Red blood cells in urine | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  Red blood cells in urine
Glomerular filtration rate | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  Glomerular filtration rate
The number of infections in the respiratory, gastrointestinal, or urinary tract | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  The number of infections in the respiratory, gastrointestinal, or urinary tract
TCM syndrome score | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  Assess the patient's clinical symptoms based on the rating scale; the higher the score, the more severe the symptoms.

OTHER OUTCOMES:
Concentration of Potassium | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  Safety indicators
electrocardiogram | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  Determine whether the patient has experienced adverse cardiac events based on the electrocardiogram
Concentration of Alanine Aminotransferase | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  Safety indicators
Concentration of Glutamic-oxaloacetic transaminase | 0 weeks, 4 weeks, 8 weeks, 12 weeks
  Security indicators
Concentration of hemoglobin | 0 weeks, 4weeks, 8 weeks, 12 weeks
  Security indicators

IPD SHARING:
Plan to Share IPD: No
Individual participant data involves the personal privacy of participants and should not be made public or shared.